CLINICAL TRIAL: NCT03494816
Title: NAXIVA- Phase II Neoadjuvant Study of Axitinib for Reducing Extent of Venous Tumour Thrombus in Clear Cell Renal Cell Cancer With Venous Invasion
Brief Title: Study of Axitinib for Reducing Extent of Venous Tumour Thrombus in Renal Cancer With Venous Invasion
Acronym: NAXIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scottish Clinical Trials Research Unit (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAXIVA; 2017-000619-17 (EudraCT Number); ISRCTN96273644 (Other: ISRCTN)
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Non-metastatic Renal Cell Carcinoma
Keywords: Neoadjuvant; Venous Tumour Thrombus; Axitinib; Mayo Classification; Nephrectomy; Thrombectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axitinib (Experimental): Axitinib - oral tablet twice daily for 8 weeks prior to surgery. Starting dose 5mg.
  Interventions: Drug: Axitinib Oral Tablet

INTERVENTIONS:
Drug: Axitinib Oral Tablet — Axitinib is an oral VEGF-receptor inhibitor. Patients are prescribed a starting dose of 5mg twice daily, escalating to 10mg in absence of dose limiting toxicities and blood pressure.
  Doses should be taken approximately 12 hours apart and patients should be instructed to take their doses at approximately the same times each day with or without food as per instruction. On clinic days only, patients will be advised to fast for 6 hours prior to their clinic visit.
  Patients should be advised to stop axitinib treatment a minimum of 36 hours and maximum of 7 days prior to week 9 nephrectomy and thrombectomy surgery.
  Dose adjustments, including dose increase or dose reduction, are permitted and should be based on clinical judgement and the guidelines provided in the protocol.
  Other Names: Inlyta; AG-013736

SUMMARY:
NAXIVA is a study of axitinib in patients with metastatic and non-metastatic renal cell carcinoma with venous invasion. Patients will be given axitinib (twice daily) for 8 weeks (at an escalated dose) and the response of the venous invasion will be assessed.

Blood, urine and tumour tissue samples will be taken prior to and during therapy to evaluate biomarkers of treatment response.

The primary objective is to assess the response of the thrombus to axitinib. Its thought that axitinib will reduce the extent of the thrombus in the inferior vena cava will reduce the extent of surgical intervention.

DETAILED DESCRIPTION:
NAXIVA is a single arm, single agent, open label, phase II feasibility study of axitinib in patients with both metastatic and non-metastatic renal cell carcinoma of clear cell histology. 20 patients will be recruited from multiple centres within the United Kingdom.

Patients who have signed informed consent and who have met all eligibility criteria will be registered into the trial.

The starting dose of axitinib will be 5mg BID and escalated to 7mg BID and then 10mg BID. A dose modification assessment will take place every 2 weeks in clinic during the 8 week pre-surgical treatment period and will be dependent on tolerability of treatment. Patients will follow an aggressive axitinib dose escalation process within the 8 week period to a maximum of 10mg BID. Patients should stop axitinib a minimum of 36 hours and a maximum of 7 days prior to surgery in week 9.

Blood, urine and tissue samples will be taken prior to and during therapy to evaluate biomarkers of treatment response. Nephrectomy and IVC tumour thrombectomy will be planned for all patients on the trial.

Response to axitinib in VTT, primary tumour and any RECIST measureable lesion will be correlated with changes in molecular markers.

Patients will be followed up in clinic at 6 & 12 weeks post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18. 2. Histologically proven clear cell RCC. 3. Immediate resection of the primary tumour considered technically possible. 4. Suitable for and willing to undergo nephrectomy (either cytoreductive or with curative intent) 4. cT3b, cT3c, cT3a (main renal vein) 5. N0, N1, or Nx 6. M0, or M1 7. ECOG performance status 0 - 1 8. Urinalysis <2+ protein. If dipstick is ≥2+ then a 24-hour urine collection should be performed and the patient may enter NAXIVA only if urinary protein is <2g per 24 hours.

9. All female patients with reproductive potential must have a negative serum or urine pregnancy test within a maximum of 14 days prior to starting trial treatment.

Exclusion Criteria:

1. For M1 patients: poor risk on Memorial Sloan Kettering Cancer Centre (MSKCC) score and deemed suitable for cytoreductive nephrectomy at time of enrolment.
2. The presence of active second malignancy. Patients will be eligible if they have adequately treated basal cell carcinoma, squamous cell skin cancer, in situ cervical cancer, stable prostate cancer or if treated with curative intent for any other cancer with no evidence of disease for 2 years. Patients with prostate cancer will be permitted entry if not receiving treatment and prostrate-specific antigen (PSA) is not rising.
3. Women who are pregnant or are breastfeeding. Female patients must be surgically sterile, be postmenopausal, or must agree to use effective contraception during the period of therapy and up to 1 week after treatment.

   Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy and for 6 months after completion of study drug (Patients who do not meet this will not be are not eligible).
4. Current signs or symptoms of severe progressive or uncontrolled hepatic, endocrine or pulmonary disease other than directly related to RCC.
5. Gastrointestinal abnormalities including: a. inability to take oral medication; b. requirement for intravenous alimentation; c. prior surgical procedures affecting absorption including total gastric resection; d. treatment for active peptic ulcer disease in the past 6 months; e. active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy; f. malabsorption syndromes.
6. Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (see section 4.4, concomitant therapy).
7. Current use, or anticipated need for treatment with, drugs that are known CYP3A4 inducers or substrates for CYP1A2 (see section 4.4, concomitant therapy).
8. Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
9. Active seizure disorder, spinal cord compression, or carcinomatous meningitis.
10. Any of the following within 12 months prior to study entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
11. Uncontrolled hypertension (>160/100 mmHg despite optimised antihypertensive treatment).
12. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
13. ALT or AST ≥ 1.5 x ULN; Bilirubin ≥ 1.5 x ULN.
14. Serum creatinine ≥ 1.5 x ULN
15. Neutrophil count < 1.0 x 109/L; platelet count < 100 x 109/L; Hb ≤ 90g/L.
16. Known severe hepatic impairment (Child-Pugh class C)
17. Known hypersensitivity to axitinib or any of its excipients. Specifically patients with hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant D Stewart, Principal Investigator — University of Cambridge
Locations (7):
- United Kingdom (7):
  - Broomfield Hospital, Chelmsford, Essex
  - Addenbrookes Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London
  - St George's Hospital, London
  - Royal Marsden, London

REFERENCES:
- [Derived] Stewart GD, Welsh SJ, Ursprung S, Gallagher FA, Jones JO, Shields J, Smith CG, Mitchell TJ, Warren AY, Bex A, Boleti E, Carruthers J, Eisen T, Fife K, Hamid A, Laird A, Leung S, Malik J, Mendichovszky IA, Mumtaz F, Oades G, Priest AN, Riddick ACP, Venugopal B, Welsh M, Riddle K, Hopcroft LEM; NAXIVA Trial Group; Jones RJ. A Phase II study of neoadjuvant axitinib for reducing the extent of venous tumour thrombus in clear cell renal cell cancer with venous invasion (NAXIVA). Br J Cancer. 2022 Oct;127(6):1051-1060. doi: 10.1038/s41416-022-01883-7. Epub 2022 Jun 23. PMID 35739300

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Axitinib - oral tablet twice daily for 8 weeks prior to surgery. Starting dose 5mg.
  Axitinib Oral Tablet: Axitinib is an oral VEGF-receptor inhibitor. Patients are prescribed a starting dose of 5mg twice daily, escalating to 10mg in absence of dose limiting toxicities and blood pressure.
  Doses should be taken approximately 12 hours apart and patients should be instructed to take their doses at approximately the same times each day with or without food as per instruction. On clinic days only, patients will be advised to fast for 6 hours prior to their clinic visit.
  Patients should be advised to stop axitinib treatment a minimum of 36 hours and maximum of 7 days prior to week 9 nephrectomy and thrombectomy surgery.
  Dose adjustments, including dose increase or dose reduction, are permitted and should be based on clinical judgement and the guidelines provided in the protocol.
Period: Overall Study
Arm/Group | Single Arm
Started | 24
Completed | 18
Not Completed | 6
Not completed — Protocol Violation | 2
Not completed — Physician Decision | 2
Not completed — Did not start trial treatment | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This is the ITT population (includes patients who did not take study drug).
Groups:
- ITT Population: The Intention-to-treat (ITT) population includes all patients registered onto the study.
Arm/Group | ITT Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 17
Age, Continuous [Median (Standard Deviation); unit: years] | 69 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Change in Mayo Classification
Description: The number and percentage of evaluable patients with a change in the Mayo Classification. A patient is defined as a responder if their Mayo level is lower at 9 weeks as compared to baseline; all other patients are defined as non-responders.
  The Mayo Classification levels are defined as follows, ordered by increasing severity:
  * Level 0: thrombus limited to the renal vein
  * Level 1: into IVC <2cm from renal vein ostium level
  * Level 2: IVC extension >2cm from renal vein ostium and below hepatic vein
  * Level 3: thrombus at the level of or above the hepatic veins but below the diaphragm
  * Level 4: thrombus extending above the diaphragm
Time Frame: Surgery and radiology assessment at week 9 in comparison to pre-axitinib assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Evaluable Patients: The evaluable population includes all patients in the ITT population who have received at least one dose of the study drug (including any patients who were enrolled in error, received study drug and were subsequently found to be ineligible).
Arm/Group | Evaluable Patients
Number analyzed (Participants) | 21
Participants
  Responder | 6
  Non-responder | 15

2. Secondary Outcome: % Patients With Change in Surgical Management
Description: The percentage of patients with a change in surgical management.
  Tumour thrombus surgical management approaches are provided below, ordered by increasing invasiveness:
  1. Thrombus - Milked back into renal vein and side clamped
  2. Infra-hepatic (IVC clamping with no liver mobilisation)
  3. Retro-hepatic (liver mobilisation and clamping below hepatic veins)
  4. Retro-hepatic (liver mobilisation and clamping above hepatic veins)
  5. Supra-hepatic (infradiaphragmatic)
  6. Supra-hepatic (supradiaphragmatic)
Time Frame: Surgical planning will be conducted at week 1 (prior to axitinib) and compared to the actual outcome at week 9.
Measure: Count of Participants; unit: Participants
Groups:
- Surgical Population: The group of evaluable patients who had surgery.
Arm/Group | Surgical Population
Number analyzed (Participants) | 17
Participants
  Improvement in control of IVC/renal vein | 6
  Deterioration in control of IVC/renal vein | 0
  No change in control of IVC/renal vein | 11

3. Secondary Outcome: Change in Venous Tumour Thrombus (VTT) Height
Description: The percentage change in VTT height. VTT height is measured as follows: if the size of the tumour is X at baseline and Y at the later timepoint, the reduction value is calculated as follows: 1-(Y/X). Therefore, positive values indicate a reduction and negative values indicate an increase.
Time Frame: Radiology assessment- The VTT height will be measured prior to axitinib and compared with the VTT height just before surgery (week 9). Both pre-axitinib and week 9 scans will be centrally reviewed by the lead NAXIVA radiologists prior to analysis.
Measure: Median (Standard Deviation); unit: percentage decrease in VTT length
Groups:
- Patients With Complete VTT Length Data at 9 Weeks: 3 patients (no 9wk scan) + 1 (ineligible) pts were not included in the assessment of this timepoint.
Arm/Group | Patients With Complete VTT Length Data at 9 Weeks
Number analyzed (Participants) | 17
percentage decrease in VTT length | 21.49 (27.60)

4. Secondary Outcome: Number of Patients With RECIST Responses
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI.
  In summary, the RECIST v1.1 response categories are:
  * Complete Response (CR): disappearance of all target lesions
  * Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions
  * Progressive Disease (PD): >=20% increase in the sum of diameters of target lesions AND an absolute increase of >5mm (or the appearence of 1+ new lesions)
  * Stable Disease (SD): neither sufficient shrinkage to for PR nor sufficient increase for PD Eisenhauer et al., 2009. Eur J Cancer; 45(2): 228-47.
Time Frame: Radiology assessment- The response rate (RECIST) will be assessed at week 9 in comparison to pre-axitinib measurements.Both pre-axitinib and week 9 scans will be centrally reviewed by the lead NAXIVA radiologists prior to analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Complete RECIST Data: 3 evaluable pts did not have the relevant data and were removed from the analysis
Arm/Group | Patients With Complete RECIST Data
Number analyzed (Participants) | 18
Participants
  Complete response | 0
  Partial response | 3
  Stable disease | 13
  Progressive disease | 2
  Non-evaluable | 0

5. Secondary Outcome: Surgical Complication Rates
Description: Morbidity will be measured according to the Clavien-Dindo classification.
  A summary of the relevant categories is as follows:
  Grade I: Any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention (inc. certain drugs, physiotherapy and wound infections that are opened at the bedside) Grade II: Complications requiring drug treatments other than those allowed for Grade I complications (inc. blood transfusion and total parenteral nutrition (TPN)) Grade III: Complications requiring surgical, endoscopic or radiological intervention (IIIa=not under general anaesthetic/IIIb=under general anaesthetic) Grade IV: Life-threatening complications (inc. CNS complications requiring intensive care, but excludes transient ischaemic attacks (TIAs)) (IVa=single-organ dysfunction (inc. dialysis)/IVb=multi-organ dysfunction) Grade V: Death of the patient Dindo et al., 2004. Ann Surg;240(2):205-13.
Time Frame: Morbidity rates will be assessed by radiology assessment using pre-axitinib and week 9 scans. Both pre-axitinib and week 9 scans will be centrally reviewed by the lead NAXIVA radiologists prior to analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Post-surgical Complications Within 30 Days: While 17 patients had surgery on this trial, only 6 patients had post-surgical complications within 30 days.
Arm/Group | Patients With Post-surgical Complications Within 30 Days
Number analyzed (Participants) | 6
Participants
  Grade I | 1
  Grade II | 3
  Grade IIIa | 0
  Grade IIIb | 0
  Grade IVa | 0
  Grade IVb | 1
  Grade V | 1

ADVERSE EVENTS:
Time Frame: Data were collected at screening, Week 1, Week 3, Week 5, Week 7, Week 9 (srugery), 6 weeks post-surgery, 12 weeks post-surgery.
Arm/Group | ITT Population
All-Cause Mortality (participants affected / at risk) | 4/24
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=24)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) — Pain at wound site
Pathological fracture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Pathological fracture to humerus
Nervous system neoplasms malignant and unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Enhancing mass on L side of cerebellum
Cardiac arrest (Cardiac disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (2)
Middle cerebral artery infarct (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (2)
Hyperglycemia (Endocrine disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=24)
Abdominal pain (Gastrointestinal disorders) | 7 (13)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7)
Asthenia (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (13)
Blood creatinine increased (Investigations) | 2 (4)
Cardiac murmur (Cardiac disorders) | 1 (2)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (14)
Deafness (Ear and labyrinth disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (14)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (15)
Dysgeusia (Nervous system disorders) | 4 (9)
Dyspepsia (Gastrointestinal disorders) | 4 (11)
Dysphonia (Psychiatric disorders) | 10 (30)
Dyspnea exertional (Cardiac disorders) | 3 (6)
Dysuria (Renal and urinary disorders) | 3 (4)
Epistaxis (Vascular disorders) | 3 (3)
Fatigue (General disorders) | 15 (47)
Flank pain (General disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (4)
Hematuria (Reproductive system and breast disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 19 (85)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Hypoesthesia (Nervous system disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (6)
Incision site pain (General disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 7 (16)
Lacrimation increased (Eye disorders) | 1 (6)
Lethargy (General disorders) | 1 (2)
Loose tooth (General disorders) | 1 (2)
Male genital examination abnormal (Investigations) | 1 (5)
Migraine (Nervous system disorders) | 1 (1)
Mucosal inflammation (General disorders) | 9 (21)
Muscular weakness (Nervous system disorders) | 6 (13)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 7 (17)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Oral candidiasis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (6)
Pain (General disorders) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (10)
Paraesthesia (Nervous system disorders) | 2 (2)
Pathological fracture (Infections and infestations) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 10 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pyrexia (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Renal pain (Renal and urinary disorders) | 1 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7)
Weight decreased (Investigations) | 6 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03494816/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03494816/SAP_001.pdf